CLINICAL TRIAL: NCT06314347
Title: Determination of Reference Values of the Figure of 8 Walk Test in Healthy Adults
Brief Title: Reference Value of Figure of 8 Walk Test
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Sponsor
Other Study IDs: gibtuipekkirmaci
Record Dates: First submitted 2024-02-21; First posted 2024-03-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Figure of 8 walk test; healthy adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Figure of 8 walk test — clinical measurement

SUMMARY:
The aim of the study is to determine the reference values of the Figure 8 Walking Test in healthy adults.

DETAILED DESCRIPTION:
The Figure 8 Walk Test is a standard clinical measurement used to evaluate advanced walking performance required in daily life. Beyond walking straight, the ability to turn is required in many situations in daily life, such as getting around a table, avoiding obstacles, and navigating the street. The validity and reliability of the figure of 8 walk test have been stated for different pathological conditions, but the normative values of the test in healthy individuals are unknown.

ELIGIBILITY:
Inclusion Criteria:

* -Above 18 years old
* No known musculoskeletal and neurological disorders
* healthy adults who are not elite or professional athletes

Exclusion Criteria:

* People with physical or cognitive impairments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Figure of 8 walk test | baseline and two weeks later
  It is a standard clinical measurement used to evaluate advanced walking performance required in daily life. In the figure-8 walking test, two cones are placed 1.5 meters apart. The individual stands in the middle of this distance. At the beginning of the test, the child walks around the first cone as fast as he can, then when he reaches the other starting point, this time he walks around the other cone. The elapsed time is recorded.

SECONDARY OUTCOMES:
Age | Baseline
  age as a years
gender | Baseline
  As a male or female
height | Baseline
  height in meters
weight | baseline
  weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katirci Kirmaci ZI, Gozacan Karabulut D, Maden C, Elpeze G, Kirmaci YS, Yildirim H, Gun Kalkin T. Determination of reference values of figure of 8 walk walk test in healthy adults. Ir J Med Sci. 2026 Jan 19. doi: 10.1007/s11845-025-04276-w. Online ahead of print. PMID 41549207